CLINICAL TRIAL: NCT00003458
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Children With Brain Tumors
Brief Title: Antineoplaston Therapy in Treating Children With Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066490; BC-BT-10 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Childhood Brain Tumors
Keywords: Anaplastic astrocytoma; Anaplastic glioma; Anaplastic oligodendroglioma; Astrocytoma; Astrocytoma pilocytic; Brain stem glioma; Craniopharyngioma; Ganglioglioma; Glioblastoma multiforme; Gliosarcoma; Medulloepithelioma; Neurocytoma; Oligodendroglioma; Oligodendroglioma-brainstem; Primitive neuroectodermal tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Craniopharyngioma; Ganglioglioma; Glioblastoma; Gliosarcoma; Neuroectodermal Tumors, Primitive; Neurocytoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Children with a brain tumor will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for childhood brain tumors provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of childhood brain tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children (> 6 months of age) with brain tumors.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which children with brain tumors receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in children with a brain tumor, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in children with a brain tumor.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (except if medically contraindicated) childhood brain tumor for which no curative therapy exists
* Measurable tumor by MRI scan performed within two weeks prior to study entry
* Tumor must be at least 5 mm

PATIENT CHARACTERISTICS:

Age:

* 6 months to 17 years

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC greater than 2000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No history of heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium
* No uncontrolled hypertension

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on stable dose for at least 1 week before study entry)

Radiation therapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Recovered from any prior surgery

Other:

* No prior antineoplaston therapy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 1996-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stanislaw R. Burzynski, Tomasz J. Janicki, Gregory S. Burzynski, Ania Marszalek. A Phase II Study of Antineoplastons A10 and AS2-1 in Children with Brain Tumors. Final Report (Protocol BT-10). Journal of Cancer Therapy 8: 173-187, 2017
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four patients were recruited between September 1996 and July 2012. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Children with a brain tumor will receive Antineoplaston therapy (Atengenal + Astugenal).
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 34
Completed | 30
Not Completed | 4
Not completed — Not evaluable | 4

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: Years] | 10.4 [0.8 to 17.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 30
Participants
  Complete Response | 1
  Partial Response | 5
  Stable Disease | 6
  Progressive Disease | 18

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 34
Percentage of participants
  6 months overall survival | 64.7
  12 months overall survival | 47.1
  24 months overall survival | 35.3
  36 months overall survival | 32.4
  48 months overall survival | 20.6
  60 months overall survival | 20.6

ADVERSE EVENTS:
Time Frame: 18 years, 5 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 21/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=34)
Hemoglobin (Blood and lymphatic system disorders) | 1 — The hemoglobin was not related to Antineoplaston therapy.
Central Venous Catheter Infection (Infections and infestations) | 2 — The central venous catheter infection was not related to Antineoplaston therapy.
Fever (General disorders) | 1 — The fever was not related to Antineoplaston therapy.
Vomiting (Gastrointestinal disorders) | 1 — The vomiting was not related to Antineoplaston therapy.
Hematoma (Skin and subcutaneous tissue disorders) | 1 — The hemotoma was not related to Antineoplaston therapy.
Hemorrhage, CNS (Nervous system disorders) | 2 — Neither of the hemorrhage, CNS were related to Antineoplaston therapy.
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1 — The infection (documented clinically): lung (pneumonia) was not related to Antineoplaston therapy.
Infection (documented clinically): Skin (cellulitis) (Infections and infestations) | 1 — The infection (documented clinically): skin (cellulitis) was not related to Antineoplaston therapy.
Hyperntremia (Investigations) | 1 — The hypernatremia was possibly related to Antineoplaston therapy.
Hydrocephalus (Nervous system disorders) | 1 — The hydrocephalus was not related to Antineoplason therapy
Neuropathy: motor (Nervous system disorders) | 1 — The neuropathy: motor was not related to Antineoplason therapy
Seizure (Nervous system disorders) | 4 — The seizures were not related to Antineoplason therapy
Somnolence/depressed level of consciousness (Nervous system disorders) | 9 — One of the somnolence/depressed level of consciousness was possibly related to Antineoplason therapy
Pain: Head/headache (Nervous system disorders) | 3 — One of the pain:headache was possibly related to Antineoplason therapy
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 — The dyspnea (shortness of breath) was not related to Antineoplaston therpy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=34)
Hemoglobin (Blood and lymphatic system disorders) | 15
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 12
Lymphopenia (Blood and lymphatic system disorders) | 10
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7
Platelets (Blood and lymphatic system disorders) | 2
Central venous catheter infection (Infections and infestations) | 7
Non-functional central venous catheter (General disorders) | 13
Thrombosis/embolism - Central venous catheter (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 24
Fever (General disorders) | 11
Rigors/chills (General disorders) | 3
Weight gain (General disorders) | 3
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Edema/Fluid retention (General disorders) | 8
Cushingoid appearance (Endocrine disorders) | 5
Anorexia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 9
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 15
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 21
Hemorrhage, CNS (Nervous system disorders) | 2
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 3
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 3
Hemorrhage, pulmonary: Nose (Respiratory, thoracic and mediastinal disorders) | 5
Petechiae (Skin and subcutaneous tissue disorders) | 3
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2
Infection (documented clinically): Mucosa (Infections and infestations) | 3
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 5
Opportunistic infection (Infections and infestations) | 4
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3
Alkaline phosphatase (Investigations) | 6
Bicarbonate, serum-low (Investigations) | 4
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 4
Hypercalcemia (Investigations) | 3
Hypercholesteremia (Investigations) | 8
Hyperglycemia (Investigations) | 13
Hypermagnesemia (Investigations) | 2
Hypernatremia (Investigations) | 12
Hypertriglyceridemia (Investigations) | 4
Hypocalcemia (Investigations) | 4
Hypoglycemia (Investigations) | 11
Hypokalemia (Investigations) | 27
Hypomagnesemia (Investigations) | 3
Hyponatremia (Investigations) | 4
Hypophosphatemia (Investigations) | 5
Proteinuria (Investigations) | 10
SGOT (Investigations) | 7
SGPT (Investigations) | 10
Uric acid, serum-high (hyperuricemia) (Investigations) | 5
Ataxia (incoordination) (Nervous system disorders) | 10
Confusion (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 6
Memory impairment (Nervous system disorders) | 2
Neuropathy: CN III Pupil, upper eyelid, extra ocular movements (Nervous system disorders) | 2
Neuropathy: cranial: CN VI Lateral deviation of eye (Nervous system disorders) | 2
Neuropathy: cranial: CN VII Motor-face; Sensory-taste (Nervous system disorders) | 2
Neuropathy: motor (Nervous system disorders) | 7
Neuropathy: sensory (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 6
Somnolence/depressed level of consciousness (Nervous system disorders) | 22
Speech impairment (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 6
Diplopia (Eye disorders) | 3
Pain: Abdomen NOS (Gastrointestinal disorders) | 6
Pain: Back (Musculoskeletal and connective tissue disorders) | 3
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 2
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 4
Pain: Head/headache (Nervous system disorders) | 21
Pain: Joint (Musculoskeletal and connective tissue disorders) | 5
Pain: Middle ear (Ear and labyrinth disorders) | 2
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 3
Pain: Neck (Musculoskeletal and connective tissue disorders) | 4
Pain: Stomach (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6
Incontinence, urinary (Renal and urinary disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No